CLINICAL TRIAL: NCT04014699
Title: Clinical Evaluation of Modified 2.2mm Microincision Phacoemulsification for Age-related Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2019KYPJ091
Record Dates: First submitted 2019-07-06; First posted 2019-07-10 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified 2.2mm micoincision (Experimental)
  Interventions: Procedure: modified 2.2mm microincision
- conventional 2.2mm microincision (Active Comparator)
  Interventions: Procedure: conventional 2.2mm microincision

INTERVENTIONS:
Procedure: modified 2.2mm microincision — enlarging the internal incision about 0.4mm for conventional 2.2mm coaxial microincision phacoemulsification
  Arms: modified 2.2mm micoincision
Procedure: conventional 2.2mm microincision — conventional 2.2mm coaxial microincision phacoemulsification
  Arms: conventional 2.2mm microincision

SUMMARY:
This study is a single-center, parallel-group, randomized controlled trial with the following objectives: to compare the incidence of post-operative descemet membrane detachment (DMD) in phacoemulsification surgery between modified and conventional 2.2mm microincision.

DETAILED DESCRIPTION:
2.2mm incision is considered an ideal incision size in phacoemulsification. However, DMD is a common and serious complication in 2.2mm microincision phacoemulsification for hard nucleus age-related cataract. DMD is originated from the incision in the operation. How to construct the appropriate incision shape and size for reducing the occurrence of DMD is an important problem to be solved urgently in phacoemulsification surgery.

The investigators found that enlarging the internal incision could increase the range of motion of surgical instruments and reduce the friction of instruments to incision. Therefore，the incidence of DMD would be reduced. The investigators developed this technique, modified 2.2mm incision, to reduce the incidence of incision-site DMD and not to increase other incision related complications.

In this trial, the investigators aim to compare modified and conventional 2.2mm incision with regard to safety and efficacy in reducing the incidence of DMD.

ELIGIBILITY:
Inclusion Criteria:

* Aged-related cataract patients between 65 and 90 years ;
* Lens nuclear opalescence grade ≥4.0 on the Lens Opacities Classification System III (LOCS III);
* Scheduled for phacoemulsification combined with intraocular lens implantation.
* The number of corneal endothelial cells > 1500cells/mm2.
* Dilated pupil diameter ≥6mm

Exclusion Criteria:

* A history of ophthalmic trauma or surgery;
* Other ophthalmic diseases such as glaucoma, uveitis, high myopia;
* Ocular factors that would make surgery challenging or dangerous, including but not limited to small pupil, shallow anterior chamber, etc.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Incidence of DMD at postoperative day 1 | postoperative day 1
  Incidence of incision-site descemet membrane detachment observed by anterior segment OCT at postoperative day 1

SECONDARY OUTCOMES:
maximal incision thickness | postoperative day 1, day 7, month 1, month 3
  maximal incision thickness measured by anterior segment OCT at postoperative day 1, day 7, month 1, month 3
surgical induced-astigmatism | postoperative day 1, day 7, month 1, month 3
  surgical induced-astigmatism was calculated at each postoperative visit using the following equation: K2 = [K1 2 + K32 -2 K1 K3 cos (2θ3 -2θ1)]1/2
the length of DMD | postoperative day 1, day 7, month 1, month 3
  the length of incision-site descemet membrane detachment measured by anterior segment OCT at postoperative day 1, day 7, month 1, month 3
Best corrected visual acuity (BCVA) | postoperative day 1, day 7, month 1, month 3
  Best corrected visual acuity (BCVA) is evaluated with an ETDRS chart at each postoperative visit
modulation transfer function (MTF)-cut off | postoperative day 1, day 7, month 1, month 3
  modulation transfer function (MTF)-cut off measured by itrace at each postoperative visit
central cornea endothelial cell loss | postoperative day 1, day 7, month 1, month 3
  Central cornea endothelial cell loss was calculated on the basis of preoperative and postoperative endothelial cell density.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, China

REFERENCES:
- [Derived] Dai Y, Liu Z, Wang W, Han X, Jin L, Chen X, Jin G, Wang L, Zhang E, Qu B, Liu J, Congdon N, He M, Luo L, Liu Y. Incidence of Incision-Related Descemet Membrane Detachment Using Phacoemulsification With Trapezoid vs Conventional 2.2-mm Clear Corneal Incision: A Randomized Clinical Trial. JAMA Ophthalmol. 2021 Nov 1;139(11):1228-1234. doi: 10.1001/jamaophthalmol.2021.4148. PMID 34647960